CLINICAL TRIAL: NCT02567734
Title: Clinical Trials of CT-guided Percutaneous Irreversible Electroporation（IRE）in the Treatment of Patients With Locally Advanced Tumors：The Safety and Efficacy Assessment
Brief Title: Clinical Trials of CT-guided Percutaneous Irreversible Electroporation（IRE）in the Treatment of Patients With Locally Advanced Tumors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Yueyong Xiao (Other)
Responsible Party: Sponsor-Investigator, Yueyong Xiao, Director of the Department, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PLAGH-YY-001
Record Dates: First submitted 2015-09-28; First posted 2015-10-05 (Estimated); Last update posted 2015-12-28 (Estimated); Status verified 2015-10

CONDITIONS: Neoplasms; Carcinoma
Keywords: irreversible electroporation; ablation; neoplasms; cancer; carcinoma; NanoKnife; Ablation Techniques
MeSH Terms: conditions — Neoplasms; Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Irreversible electroporation (Experimental): In this group，eligible patients were selected to receive the CT-guided percutaneous irreversible electroporation ablation.
  Interventions: Procedure: CT-guided percutaneous irreversible electroporation

INTERVENTIONS:
Procedure: CT-guided percutaneous irreversible electroporation — Patients undergo the irreversible electroporation ablation that induce protracted cell death by apoptosis through cell membrane perforation.All these procedures will be performed under the guide of Big bore multislice spiral CT scanning system.
  Other Names: NanoKnife

SUMMARY:
Irreversible electroporation (IRE) is an emerging nonthermal focal ablation technique that uses a series of short but intense electric pulses delivered by NanoKnife generator through paired electrodes into a targeted region of tissue, inducing the cells death by apoptosis through irreversibly disrupting cellular membrane integrity. This study aimed to investigate the safety and efficacy of CT-guided percutaneous irreversible electroporation（IRE） in the treatment of patients with locally advanced tumors in different anatomical position.

DETAILED DESCRIPTION:
This study is a multicenter, open-label trial that aimed to evaluate the safety and efficacy of CT-guided percutaneous irreversible electroporation（IRE）in the treatment of patients with locally advanced tumors. Investigators will screen eligible patients and examine them by imaging tests as well as serological examination before and after the IRE procedures to assess the result with the size，blood supply，metabolism of tumors，the change of blood test and treatment-related complications. Big bore multislice spiral CT with thickness 5 cm, 120kilovolt，and 250milliampere，ECG-gated device and anesthesia monitoring equipment were selected during these procedures. Imaging (performed by contrast enhanced CT scan) and serological follow-up was at postoperative day 3 and 1，3，6，12months. The primary endpoint is the effective rate of IRE，and the secondary endpoint is 1-year survival rate and the frequency of adverse events. The response of irreversible electroporation ablation will be assessed according to the different evaluation criterions based on Response Evaluation Criteria in Solid Tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed locally advanced solid tumor.
2. Unresectable tumors or the patient refused surgical therapy.
3. Patients in good health conditions can receive general anesthesia.
4. Patients with good compliance can cooperate with doctors for related tests and the regular follow-up.

Exclusion Criteria:

1. Targeted tissues that metallic wallstents or metallics were implanted.
2. With heart pacemaker or be allergic to contrast medium that can not have related imaging examinations.
3. With bleeding and psychiatric disorders.
4. Severe arrhythmia.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-12 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
effective rate of IRE ablation | up to 12 months after the procedures
  The procedure-related result will be assess by the size，blood supply，metabolism of the tumors. The changes of blood test are also considerable.

SECONDARY OUTCOMES:
1-year survival rates | up to 12 months after the procedures
complication rate | During the procedure or up to 12 months after the ablation procedure
  the frequency of adverse events，including early and late complications

CONTACTS AND LOCATIONS:
Overall Officials: Yueyong Xiao, Principal Investigator — The Chinese PLA General Hospital
Locations (1):
- The Chinese PLA General Hospital, Beijing, China